CLINICAL TRIAL: NCT00937053
Title: The Effect of Maintaining a Higher Haemoglobin Level on Neutropenia Duration After Bone Marrow Transplantation in Children.
Brief Title: Maintaining a Higher Level of Haemoglobin: Effect on the White Cells After Bone Marrow Transplantation in Children.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 3 unexpected Serious Adverse Events (veno-occlusive disease (VOD))
Sponsor: St. Justine's Hospital (Other)
Collaborators: Nancy Robitaille, MD (Unknown)
Responsible Party: Michel Duval, CHU Sainte-Justine, Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9967
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2009-05

CONDITIONS: Neutropenia
Keywords: Neutropenia; Transfusions; Hemoglobin; Bone marrow transplant; Hematopoietic stem cell transplant
MeSH Terms: conditions — Neutropenia | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemoglobin below 120 g/dL (Experimental)
  Interventions: Other: Transfusion level 120 g/dL; Other: Platelet transfusion
- Hemoglobin below 70 g/dL (Active Comparator)
  Interventions: Other: Transfusion level 70 g/dL; Other: Platelet transfusion

INTERVENTIONS:
Other: Transfusion level 120 g/dL — Patients whose hemoglobin falls below 120 g/dL will be transfused with red cells within 24 hours.
  Arms: Hemoglobin below 120 g/dL
Other: Transfusion level 70 g/dL — Patients whose hemoglobin falls below 70 g/dL will be transfused with red cells within 24 hours
  Arms: Hemoglobin below 70 g/dL
Other: Platelet transfusion — Patients whose platelets fall below 10 x 10*9 will be transfused with platelets

SUMMARY:
The purpose of this study is to determine if maintaining a high hemoglobin level in children that underwent bone marrow transplant will accelerate the neutrophil recovery.

DETAILED DESCRIPTION:
The investigators know that children requiring bone marrow transplant need to first go through a myeloablative regimen, which induces a neutropenia. The length of the neutropenia has an incidence on the risk of contracting bacterial and fungal infections that could be lethal. It is then important to find ways to accelerate the neutrophil recovery, so patient survival can be improved.

Studies conducted in the '70s and '80s suggested that if the hemoglobin level could be kept at a higher level, then the neutrophil recovery would be accelerated. Other studies also support the hypothesis that if the stem cells do not need to produce red cells because these are being supplied through transfusions, then the stem cells would differentiate into non-erythroid cell lines.

As of now, for patients undergoing a bone marrow transplant, it is standard practice to transfuse with red cells based on the condition of the patient or if the hemoglobin level falls below 70 g/L. Hematopoietic growth factors have been used to increase the speed of the neutrophil recovery, but studies conducted so far do not demonstrate that mortality and length of hospitalization have been reduced by the specific use of G-CSF. In more recent studies, these agents have been shown to also have negative effects, such as delayed platelet recovery and impaired immune recovery. In addition, the prophylactic use of G-CSF was also associated with graft-versus-host disease, treatment-related mortality and death.

In conclusion, this study will determine if maintaining a higher hemoglobin level has an effect on the neutrophil recovery after allogenic bone marrow transplantation in children.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 1 year of age and 18 years of age at the time of transplantation (18 years is the upper limit of childhood in CIBMTR definitions)
2. Patients planned to undergo a related or unrelated allogeneic bone marrow transplant for a malignant or benign disease (except for sickle cell disease)
3. Conditioning regimen must be myeloablative, i.e. include busulfan greater or equal to 12 mg/kg or Total Body Irradiation greater or equal to 10 Gy, except for patients with acquired severe aplastic anemia
4. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before enrolment in the trial
5. Patient must agree to receive blood transfusion
6. Patient (or their legal guardians) must sign an Informed consent Form

Exclusion Criteria:

1. Patients receiving autologous bone marrow transplant, cord blood transplant or peripheral stem cell transplant
2. Sickle cell disease (since higher hemoglobin level increases blood viscosity and puts these patients at risk for stroke)
3. Hematopoietic growth factor (G-CSF, GM-CSF, stem cell factor, erythropoietin) planned before transplantation (post-transplant decision of hematopoietic growth factors administration as required by the patient's condition will be accepted)
4. Presence of an allo-antibody directed against red blood cells

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil engraftment (defined as the time from transplantation to the first of three consecutive days with a neutrophil count > 0,5 x 109/L, as used in the International Bone Marrow Transplant Registry (IBMTR) criteria). | First 100 days post HSCT

SECONDARY OUTCOMES:
Time to platelet engraftment (defined as the time from transplantation to the first of three consecutive days with a platelet count > 20 x 109/L, without platelet transfusion 7 days prior (IBMTR criteria)). | First 100 days post HSCT
Transfusions given (red cells and platelets) | First 100 days post HSCT
Hospitalization length | 2 years
Immune reconstitution (lymphoid subsets) | First 100 days post HSCT
Overall survival | 5 years
Graft vs host disease (GVHD) | 2 years
Treatment-related mortality (death without relapse) | 2 years
Relapse | 2 years
Chimerism | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel Duval, MD, Principal Investigator — St. Justine's Hospital; Nancy Robitaille, MD, Principal Investigator — St. Justine's Hospital
Locations (5):
- Canada (5):
  - Souther Alberta Children's Cancer Care Program, Calgary, Calgary, Alberta
  - Pediatric Bone Marrow Transplant Unit, British Columbia Children's Hospital, Vancouver, British Columbia
  - Section of Blood and Marrow Transplant, The Hospital for Sick Children, Toronto, Ontario
  - Hematopoietic Stem Cell Transplantation Program, Sainte-Justine Hospital, Montreal, Quebec
  - Department of Hematology, The Montreal Children's Hospital, Montreal, Quebec